CLINICAL TRIAL: NCT06061380
Title: Challenges and Management of Post-intubation Tracheal Stenosis: A Case Report and Literature Review
Brief Title: Challenges and Management of Post-intubation Tracheal Stenosis
Status: Completed | Type: Observational
Sponsor: Wollo University (Other)
Responsible Party: Principal Investigator, Aynalem Befkadu Woldemichael, Principal Investigator, Wollo University
Other Study IDs: 458840
Record Dates: First submitted 2023-05-14; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Tracheal Stenosis
MeSH Terms: conditions — Tracheal Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervation taken

SUMMARY:
Management of a "difficult airway" remains one of the most relevant and challenging tasks for anesthesiologists and pulmonary physicians. Tracheal stenosis is not common but serious complication of prolonged intubation and tracheostomy patients. The incidence of stenosis is very low if intubation lasts less than a week and patients may be asymptomatic for a long time. On presentation, tracheal stenosis may be mistaken for asthma with dyspnea and stridor. The choice of treatment depends on the site, grade, and length of stenosis, as well as on patient comorbidities, history of previous interventions, and the expertise of the surgical team. In this case report the investigators wanted to present a case of a 25-year-old female with post-intubation tracheal stenosis who was intubated for the management of severe preeclampsia.

DETAILED DESCRIPTION:
Trachea stenosis is a rare but life-threatening condition and is caused by congenital problems, post-intubation injury, trauma from surgery, tracheal tumor and compression of the trachea by tumor, or accidents, inhalation injuries or inflammatory diseases such as Wegener's granulomatosis, sarcoidosis, or systemic lupus erythematous. The investigator would like to report tracheal stenosis secondary to prolonged intubation

Case presentation

A 25-year-old female patient (height, 150 cm; weight, 50kg; body mass index, 20kg/m2) was referred to Minilik referral hospital from Debrebirhan referral hospital with a history of prolonged intubation (7 days), following severe eclampsia and uncontrolled seizure. She gives birth through spontaneous vaginal delivery in a local health care center and she doesn't know that she was preeclamptic before delivery and develops seizures after delivery so she was admitted to ICU to control her airway and stayed on a mechanical ventilator for 7 days. After extubation, she develops shortness of breath and difficulty talking. During the preoperative visit, the investigator found her on a face mask with a flow rate of 2 l/mint. She has difficulty in breathing and a dry cough associated with the stenosis but no fever or other symptoms of acute infection. Hypertension was controlled and no complications were associated with it. She had no family history of disease or any notable medical conditions. On physical examination, she has normal findings with stable vital signs of RR =21, PR =80, and BP =140/90. A three-dimensional CT scan of the neck shows trachea stenosis 14mm in length with 5mm in thickness of the wall at the level of the sternal notch. Chest CT scan also reveals tracheal stenosis at the thoracic inlet. Her complete blood profile, kidney function test, liver function test, clotting parameters, and electrocardiogram were within normal limits.

On the day of surgery, the patient was taken to the operation theatre while she was on face mask O2 and written informed consent was taken. Two wide-bore peripheral lines were secured and the patient was premeditated with dexamethasone 8mg in OT. Then the team transferred her to the OR quickly and applied the minimum standard monitoring (SpO2, non-invasive BP, ECG, and ETCO2 monitoring) in a sitting position while she was on nasal oxygen. 50 mg peptide was administered. Difficult airway was anticipated and a difficult airway cart was kept ready. Small size cuffed tubes up to 4mm ID were arranged. The patient was pre-oxygenated in a sitting position with 3 VC breathing and an induction dose of propofol (100mg) was given and halothane opened at 3% concentration. 2mg/kg of IV lidocaine was given and as anesthesia deepened laryngoscopy started. During direct laryngoscopy, the cord is visible posteriorly with a good view and intubation was tried with a cuffed tube 6.0 mm ID. The tube passed the glottis but unable to advance below it and immediately this tube changed to 5.0 mm but it was failed. Finally, a 4.0 mm ID tube was inserted by rotating side to side gently and the cuff was inflated to prevent any gas leakage, and the tube was secured at the 20 cm mark. There was significant resistance in the breathing bag so the patient was ventilated by decreasing tidal volume and increasing the rate for keeping Etco2 between 30- 35. Due to the manipulation and preexisting hypertension, BP was raised up to 200/115 so the investigator administered 5 mg hydralazine and 100mg hydrocortisone for the manipulation. Anaesthesia was maintained with Oxygen and Isoflurane with an injection of vecuronium intermittently. After securing the airway and proper positioning surgery was started. IV fluid was warmed and the required fluid amount was run in both hands. When the surgeon reached the stenosis part they inserted another sterile 6.0 mm tube below the stenosis. the surgeon's anastomosis of the remaining part.

Mid sternotomy was done and the stenosed segment was opened, a second cuffed ETT of 6.0 mm ID was passed through the distal tracheal segment (below the stenosis) by the surgeon. The circuit was disconnected from the first endotracheal tube and new sterile ventilator tubing was connected to the second endotracheal tube to continue ventilation. Bilateral air entry confirmed the tube was secured by suture applied by surgeons the cuff inflated to minimize the air leakage, and the patient was ventilated. After resection of the stenosis part, the oral 4.0mm tube was changed by a 6.0 mm tube. The cuff was inflated to prevent a gas leak. Bilateral equal chest movement was visualized. Surgery was kept continued and 1 unit of blood was given after the patient had her allowable blood loss. After completion of surgery and the appearance of adequate respiratory efforts, 1mg atropine and 2.5 mg neostigmine were given for reversal, and the patient was shifted to ICU with an endotracheal tube in situ on spontaneous respiration. The patient was extubated when she became awake with a respiratory rate of 20, HR=89, BP=128/84 adequate breathing.

H story summary History of present illness: shortness of breathing due to tracheal stenosis General condition: Awake, Alert, and Oriented, wt. 50, Ht. 150cm Medications: hydrocortisone 100mg IV BID Allergies: Not Known Drug Allergy Past Medical History: eclampsia Physical Exam: V/S: within the normal limit for age; BMI= 20 HEENT: pink conjunctive, tonsillar enlargement, otherwise normal Airway exam: TMJ: free/mobile Mallampati class II, stridor Pulmonary: Clear to auscultation and percussion, bilateral air entry with equal breath sound, no wheezing CVS: s1 & s2 well heard + no murmur or gallop Investigation: Hgb./Hct.: 12.3/39 BG: O +ve, PT=12 seconds (5-14) INR: 1.2, Platelets: 283,000, ECG normal Assessment: ASA II + tracheal stenosis + preeclampsia + fit for anesthesia

ELIGIBILITY:
Inclusion Criteria:

* Cases with tracheal stenosis caused by only prolonged intubation
* Female

Exclusion Criteria:

* Any tracheal stenosis caused by trauma, mass compression
* Being male

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A mother developing post-intubation tracheal stenosis
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2021-01-23 (Actual); Primary Completion 2021-01-24 (Actual); Study Completion 2021-01-24 (Actual)

PRIMARY OUTCOMES:
post-intubation tracheal stenosis | the patient was follwed for 1 wk
  The severity of tracheal stenosis was based on Cotton criteria confirmed by a Computerized tomography (CT) scan and the size of the tube that passed through it. If the Tracheal diameter is> 8 mm but symptomatic mild, 5-8 mm moderate, and <5 mm severe, and the effect of the severe tracheal stenosis was observed on anesthesia position, tracheal intubation technique, tube size that would challenge anesthesia management is reported

CONTACTS AND LOCATIONS:
Overall Officials: Aynalem Bk Woldemichael, MSC, Principal Investigator — Wollo Universty
Locations (1):
- Dessie comprehensive specilized hospital, Dessie, Amhara, Ethiopia

IPD SHARING:
Plan to Share IPD: No